CLINICAL TRIAL: NCT04552093
Title: Hepatic Arterial Infusion PUMP Chemotherapy Combined With systemIc chemoTherapy for Potentially Resectable Colorectal Liver Metastases: The PUMP-IT Study.
Brief Title: Hepatic Arterial Infusion Pump Chemotherapy Combined With Systemic Chemotherapy (PUMP-IT)
Acronym: PUMP-IT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19PIT; NL70112.031.19 (Registry Identifier: Registry ID: CCMO); 2019-003260-44 (EudraCT Number)
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasms
Keywords: Hepatic artery infusion pump; Colorectal liver metastases; FUDR; Floxuridine; CRLM
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Floxuridine

STUDY DESIGN:
Intervention Model Description: Patients with potentially resectable (i.e. unresectable or upfront resectable with an indication for upfront systemic therapy) will receive hepatic artery infusion pump chemotherapy, consisting of floxuridine (FUDR), combined with standard of care systemic therapy (FOLFOX or FOLFIRI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Colorectal liver metastases (Experimental): Patients with potentially resectable colorectal liver metastases will undergo hepatic artery infusion pump placement. Subsequent hepatic artery infusion of floxuridine via the HAIP as well as standard of care Dutch systemic chemotherapy (FOLFOX or FOLRIRI) will be administered in a combined chemotherapy schedule.
  Interventions: Drug: Floxuridine; Device: Tricumed IP2000V infusion pump

INTERVENTIONS:
Drug: Floxuridine — Administration of intra-arterial floxuridine via the HAIP (HAIP chemotherapy) to the liver with concomitant Dutch standard of care systemic FOLFOX (5-FU, leucovorin and oxaliplatin) or FOLFIRI (5-FU, leucovorin and irinotecan).
  Other Names: FUDR
Device: Tricumed IP2000V infusion pump — Surgical implantation of hepatic artery infusion pump (HAIP) followed by administration of the combined chemotherapy (HAIP and systemic).

SUMMARY:
The PUMP-IT study is designed to prove the feasibility of HAIP chemotherapy with concomitant standard systemic chemotherapy (FOLFOX and FOLFIRI) in the Netherlands. This study will include patients with both unresectable CRLM and resectable CRLM with an indication for upfront systemic therapy (further referred to as potentially resectable CRLM), without extrahepatic metastases. The study will be performed in two tertiary referral centers in the Netherlands.

DETAILED DESCRIPTION:
RATIONALE - Colorectal cancer (CRC) is the third most common cancer with an annual incidence of 14.000 patients in the Netherlands. Of all patients with metastases, 32% have isolated colorectal liver metastases (CRLM). Local treatment of CRLM, i.e. resection, ablation and/or stereotactic radiotherapy, is the only potentially curative option. Unfortunately over 75% of these patients have CRLM which are (initially) not suitable for such local treatment.

Current treatment of unresectable CRLM includes subsequent lines of systemic (chemo)therapy aiming to convert the CRLM from an unresectable to a resectable or local treatable state in order to prolong survival. Conversion rates of modern first line systemic chemotherapeutic regimens, as described in multiple retrospective studies with highly selected patients, are observed in 10-76% of patients, resulting in a 5-year survival of 33-43% after conversion. Patients with progressive disease on first line therapy are offered second line systemic therapy. Conversion during second line systemic therapy is rare and described in only 7-13.5% of patients. These patients have a poor prognosis with a median OS of approximately 10-15 months. However, overall survival (OS) of patients undergoing local treatment after conversion on second line systemic therapy is comparable to what is observed after conversion on first line systemic therapy.

Hepatic arterial infusion pump (HAIP) can deliver high-dose regional chemotherapy to the CRLM using their unique arterial blood supply. Floxuridine is used for HAIP chemotherapy because of the advantages of having a half-life of ten minutes, a 95% first-pass effect and allowing high intrahepatic dosing resulting in increased hepatic exposure by a factor 400, with minimal systemic exposure (e.g. complications). These specific properties of HAIP chemotherapy make it possible to combine high-dose local HAIP therapy with standard of care systemic therapy.

Several single center studies from Memorial Sloan Kettering Cancer Center (MSKCC) (New York, USA) have shown high response rates with HAIP chemotherapy in combination with systemic therapy for unresectable CRLM. Conversion to resection of the initially unresectable CRLM have been observed in up to 57% of chemo-naïve patients and in 20%-38% of patients with prior systemic therapy treated with the combination of HAIP and systemic therapy. Irrespective of conversion, the combined therapy resulted in a median OS of 50.8-76.6 months and a 5-year OS of 51.9% for chemo-naïve patients. The median and 5-year OS was 27.7-35 months and 27.9%, respectively, for patients who have been treated with systemic therapy before.

Although these results are impressive, they come from a single center and have not yet been confirmed elsewhere. Most important reasons were the technically challenging surgical procedure of HAIP implantation and the need for stringent monitoring and specific management of HAIP chemotherapy requiring a highly skilled multidisciplinary treatment team.

A study investigating combined treatment is required to prove feasibility in a multicenter setting outside MSKCC before a multicenter randomized phase III trial can be initiated in the Netherlands.

STUDY DESIGN - All eligible patients who signed informed consent (registration) and meet all inclusion criteria (inclusion) will undergo surgical HAIP implantation. HAIP function is evaluated with a perfusion test during surgery and postoperatively before starting drug treatment. Start of combined HAIP chemotherapy and systemic chemotherapy is aimed within 6 weeks postoperatively. Clinical and laboratory evaluations and chemotherapy administration are scheduled every two weeks. Response evaluations will be conducted with CT thorax/abdomen and CEA measurement every 2 HAIP cycles (every 4 systemic chemotherapy cycles) during combined therapy.

The combined therapy cycles are continued until disease progression, severe toxicity, CRLM conversion to surgical local treatment or patients withdrawal. After HAIP chemotherapy discontinuation, treatment and/or follow-up are according to standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ECOG performance status 0 or 1.
* Life expectancy of at least 12 weeks.
* Histologically confirmed CRC.
* Indication for first or second line systemic therapy, confirmed in a multidisciplinary meeting.
* Potentially resectable (i.e. unresectable and upfront resectable CRLM with indication for neoadjuvant systemic therapy), confirmed in a multidisciplinary meeting and radio-logically on (PET) CT thorax/abdomen and/or MRI obtained ≤ 4 weeks prior to regis-tration.
* Positioning of a catheter for HAIP chemotherapy is technically feasible confirmed in the multidisciplinary liver meeting based on imaging. The default site for the catheter insertion is the gastroduodenal artery (GDA). Accessory or aberrant hepatic arteries are no contra-indication for catheter implantation. The GDA should have at least one branch to the liver, accessory or aberrant hepatic arteries should be ligated to allow for cross perfusion to the entire liver through intrahepatic shunts.
* Indication and eligibility for abdominal surgery confirmed in a multidisciplinary meeting, e.g. primary tumour resection, stoma revision/reversal and diagnostic surgery.
* In case of primary tumour in situ: tumour should be (potentially) resectable, confirmed in a multidisciplinary meeting.
* Adequate bone marrow, liver and renal function as assessed by the following labora-tory requirements to be conducted within 15 days prior to inclusion.

  * Hb ≥ 5.5 mmol/L
  * Absolute neutrophil count (ANC) ≥1.5 * 109/L
  * Platelets ≥100 * 109/L
  * Total bilirubin < 1.5 mg/dL
  * ASAT ≤ 5 * times the upper limit of normal (ULN)
  * ALAT ≤ 5 * ULN
  * Alkaline phosphatase ≤ 5 * ULN
  * (estimated) glomerular filtration rate (eGFR) > 45 ml/min.
* Before patient registration, written informed consent must be given and signed according to ICH-GCP, and national/local regulations.

Exclusion Criteria:

* Extrahepatic metastases. Confirmed with CT thorax/abdomen obtained ≤ 4 weeks prior to registration. Patients with small (≤ 1 cm) extrahepatic lesions that are not clearly suspicious of metastases are eligible.
* Prior hepatic radiation, resection (other than biopsy), or ablation.
* Concurrent malignancies that interfere with the planned study treatment or the prognosis of CRLM.
* Participation in other clinical trials interfering with the study treatment as judged by the treating physician.
* Dihydropyrimidine dehydrogenasedeficiency (DPD deficiency).
* Pregnant or lactating women.
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.
* Organ allografts requiring immunosuppressive therapy.
* Serious, non-healing wound, ulcer, or bone fracture.
* Chronic treatment with corticosteroids (dose of ≥ 10 mg/day methylprednisolone equiv-alent excluding inhaled steroids).
* Serious infections (uncontrolled or requiring treatment).
* History of psychiatric disability judged by the investigator to potentially hamper compliance with the study protocol and follow-up schedule.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of 2 combined chemotherapy cycles (feasibility) | Approximately 4 months after patient inclusion
  The percentage of patients that complete two cycles of combined chemotherapy (HAIP chemotherapy and systemic therapy) after being scheduled for surgical implantation.

SECONDARY OUTCOMES:
Safety: Postoperative complications | 90 days after surgery
  Surgical complications will be defined according to Clavien-Dindo surgical complications score. Complications of Clavien-Dindo grade 3 or higher are recorded for the first 90 days after surgery. Postoperative complications include those related to the HAIP implantation. Postoperative mortality is defined as any death during hospitalization or within 90 days from surgery.
Safety: Drug treatment toxicity | 1.5 year
  Toxicity grade 3 or higher will be recorded from the time of study inclusion according to the CTCAE criteria.
Safety: Other adverse events | 1.5 year
  Treatment related serious adverse events (SAE) and adverse events (AE) of grade 3 or higher will be collected continuously from the time of study inclusion until the end of combined chemotherapy. AE are followed up until the event is either resolved or adequately explained, even after the patient has completed his/her study treatment. Nature and duration of any hospitalization, treatment of any AE, and nature and duration of any outpatient care will be recorded.
Response rate colorectal liver metastases (CRLM) | 8 months after patient registration
  Response rates of CRLM will be measured according to RECIST criteria
Progression free survival (PFS) | 1.5 year
  PFS will be defined from inclusion date until disease progression.
Overall survival (OS) | 1.5 year
  OS will be defined from inclusion date until death.
Conversion rate colorectal liver metastases (CRLM) | 8 months after patient inclusion
  Conversion rate is defined as the percentage of patients in whom CRLM convert from an unresectable to a resectable state and undergo surgical treatment with curative intent. Possibility of local treatment is at the discretion of the multidisciplinary liver panel.

OTHER OUTCOMES:
Quality of life assessment | 8 months after patient inclusion
  The quality of life will be examined with validated questionnaires (EORTC QLQ-C30 & EQ-5D-3L).

CONTACTS AND LOCATIONS:
Overall Officials: Koert FD Kuhlmann, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, Netherlands

REFERENCES:
- [Derived] Krul MF, Kok NFM, Osmani H, Buisman FE, Groot Koerkamp B, Grunhagen DJ, Verhoef C, Mostert B, Snaebjornsson P, Westerink B, Klompenhouwer EG, Donswijk ML, Ruers TJM, Douma JAJ, van Blijderveen N, Kingham TP, D'Angelica MI, Kemeny NE, Bolhuis K, Buffart TE, Kuhlmann KFD. Hepatic arterial infusion pump chemotherapy combined with systemic chemotherapy for borderline resectable and unresectable colorectal liver metastases: phase II feasibility study. Br J Surg. 2024 Apr 3;111(4):znae089. doi: 10.1093/bjs/znae089. PMID 38608150